CLINICAL TRIAL: NCT05911178
Title: Impact of Microglial Activation on Synaptic Density in Alzheimer's Disease
Acronym: GliSyn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: D23-P006
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: Neuroinflammation; Microglial activation; Synaptic density; Tau pathology; Peripheral immunity
MeSH Terms: conditions — Alzheimer Disease; Neuroinflammatory Diseases | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Intervention Model Description: Early and late onset AD subjects, matched to controls for age and education level, will be followed up for two years, allowing both longitudinal and cross-sectional comparisons.
Masking Description: This is a non-randomized, open label study including three groups; early onset AD, late onset AD, healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Onset Alzheimer's Disease (EOAD) (Experimental): Patients who have been diagnosed with AD according to clinical and biomarker criteria. Early onset AD is considered as having an age of onset of symptoms younger than 65 years.
  Age of onset ≤ 65 years
  Interventions: Radiation: [11C]-UCB-J; Radiation: [18F]-DPA-714; Radiation: [18F]-RO-948
- Late Onset Alzheimer's Disease (LOAD) (Experimental): Patients who have been diagnosed with AD according to clinical and biomarker criteria. Late onset AD is considered as having an age of onset of symptoms older than 65 years.
  Age of onset > 65 years
  Interventions: Radiation: [11C]-UCB-J; Radiation: [18F]-DPA-714; Radiation: [18F]-RO-948
- Controls (Experimental): Healthy control subjects will be matched to patients for age and education level.
  Interventions: Radiation: [11C]-UCB-J; Radiation: [18F]-DPA-714; Radiation: [18F]-RO-948; Radiation: [11C]-PiB

INTERVENTIONS:
Radiation: [11C]-UCB-J — PET tracer binding to "SV2A" protein, used to study synaptic vesicle density.
Radiation: [18F]-DPA-714 — PET tracer binding to "TSPO" protein, used to study microglial activation.
Radiation: [18F]-RO-948 — PET tracer binding to "tau" protein, used to study the topography of tau deposition.
Radiation: [11C]-PiB — PET tracer binding to Aβ40 and Aβ42 fibrils and insoluble plaques containing the aforementioned Aß peptides, used to study the topography of amyloid deposition.
  Arms: Controls

SUMMARY:
This study aims to analyse, in vivo, the interplay between microglial activation and tau pathology in Alzheimer's disease (AD) using [18F]-DPA-714 and [18F]-Ro948 tracers by Position Emission Tomography (PET), and their consequences on synaptic density using [11C]-UCB-J, a recent PET radioligand.

By coupling advanced neuroimaging techniques in AD patients, while comparing them to controls, we will be able to study, for the first time in humans, the interaction between neuroinflammation, tau pathology, synaptic density, and their impact on AD progression. Joint analyses of peripheral immune biomarkers, carried out as a secondary objective, will further aim at defining peripheral correlates of this interplay.

Overall, we aim to refine AD subgroup classification in order to improve and to refine the design of new therapeutic trials.

DETAILED DESCRIPTION:
The present study aims to reevaluate the interplay between microglial activation, tau pathology, and synaptic density. It is an interventional, comparative, controlled, non-randomized study in which AD patients will be matched to controls. In order to better our current understanding of pathophysiological processes of neuroinflammation in AD, we will analyze regional microglial activation, cortical tau deposition, and synaptic dysfunction by employing multiple PET radioligands and MRI. The hybrid images will be acquired at baseline and at two years.

This study design opens the door to a multimodal study; first transversal (by determining whether the level and the extent of DPA-714 binding are associated with synaptic loss and tau deposition) then longitudinal (after a two-year follow-up based on PET/MRI, cognitive and clinical assessment and peripheral immune biomarkers). By using PET imaging at baseline and at two years, we will investigate the neuroinflammation dynamics in sporadic AD and its consequences on neurodegenerative biomarkers as well as its clinical repercussions.

Conservative diagnosis criteria based on clinical and CSF biomarkers have been established to avoid risks of misdiagnosis for the patients. The controls will undergo, at inclusion, an additional PiB-PET imaging to avoid bias and to identify amyloid positive controls.

A complete clinical and cognitive evaluation will accompany the image acquisition at baseline. The subjects will be followed up clinically at one year. At two years, another set of PET/MRIs will be performed as well as a cognitive evaluation. The image acquisitions will be planned within 6 months of each clinical visit at baseline and at two years.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Adult (older than 18 years)
* Women old enough to procreate under effective contraception
* Signed consent
* Absence of general or systemic disorders that may interfere with cognition.

Inclusion criteria for EOAD and LOAD patients:

* Progressive amnestic syndrome, associated or not with other cognitive impairments,
* CDR = 0.5 or 1
* Absence of general or systemic disorders that may interfere with cognition or PET imaging analysis,
* Absence of brain lesions as determined by MRI carried out within the framework of usual care.
* Presence of CSF biomarkers profile suggestive of AD

Inclusion criteria for controls:

* absence of subjective problems with memory and normal scores on the MMSE (MMSE > 27) with no more than one word missing.
* older than 50 years old.
* Scores on the Free and Cued Selective Reminding Test (FCSRT) of >25 for free recall and >44 for total recall.
* absence of general or systemic disorders that may interfere with cognition at follow-up.

Controls will be matched to AD patients for age and education level.

Exclusion Criteria:

* Subject with a psychiatric evolutionary and/or poorly checked pathology (left to the judgement of the investigator).
* Subject with a grave, severe or unstable pathology (left to the judgement of the investigator) the nature of which can interfere with the variables of evaluation.
* Current auto-immune disease
* Subject presenting contraindications to the 3T MRI
* Known or supposed histories (≤5 years) of severe alcoholism or misuse of drugs
* Vascular, inflammatory or expansive, visible lesion in the MRI which can interfere on the criteria of diagnosis.
* No health insurance
* Pregnant, breast-feeding woman or planning a pregnancy in two years of follow-up.
* Diagnosis or history of other possible etiology of dementia, including but not limited to other neurodegenerative disorders.
* Person placed under the protection of justice
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2028-02-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Change in regional microglial activation and tau pathology from baseline at 24 months | 24 months
  The first primary endpoint will be evaluated and compared to baseline across all participants (patients and controls). The microglial activation and tau pathology will be measured respectively with [18F]-DPA-714 and [18F]-RO-948 binding rate at baseline and again at 24 months. The change will be calculated by comparing the baseline and 24-month uptake ratios.
Change in regional synaptic density from baseline at 24 months | 24 months
  The second primary endpoint will be evaluated and compared to baseline across all participants (patients and controls). The synaptic density will be measured with [11C]-UCB-J. We hypothesize that both tau pathology and microglial activation will modulate regional synaptic density, which is responsible for clinical symptoms. The change will be calculated by comparing the baseline and 24-month uptake ratios.

SECONDARY OUTCOMES:
Change in neuroimmune reaction as assessed by [18F]-DPA-714 PET global cortical index and regional cortical binding at baseline and at 24 months across all participants | 24 months
  Global and regional cortical [18F]-DPA-714 uptake ratio.
Incidence of novel peripheral and CSF immune biomarkers across all participants at baseline, at 1 year, and at 2 years | 24 months
  Peripheral and CSF immune biomarkers will be identified by broad spectrum immunophenotyping in order to determine, if any, novel biological markers of prognosis on disease evolution over 1 and 2 years of follow-up.
Rate of clinical disease progression as impacted by global and regional tau deposition at baseline, at 1 years, and at 2 years | 24 months
  Clinical presentation of symptoms will be mainly evaluated by the changes in MMSE (total score out of 30) and CDR (total score out of 3) scores. And it will be compared with the topography of tau deposition (measured by [18F]-RO-948) for each patient.
Rate of clinical disease progression as impacted by global and regional synaptic density at baseline, at 1 years, and at 2 years | 24 months
  Clinical presentation of symptoms will be mainly evaluated by the changes in MMSE (total score out of 30) and CDR (total score out of 3) scores. And it will be compared with the synaptic density (measured by [11C]-UCB-J) for each patient.
Comparison of the rate of central and systemic inflammation between sporadic AD groups assessed by [18F]-DPA-714 PET global cortical index and regional cortical binding at baseline and at 24 months | 24 months
  Global and regional cortical [18F]-DPA-714 uptake ratio across the patient groups.
Correlation of the rate of clinical decline with the rate of PET tracer uptake increase at 24 months across all patients. | 24 months
  Global and regional uptake ratios will be compared to the rate of clinical decline as assessed by changes in MMSE (x/30) and CDR (x/3) scores
Correlation between the rate of clinical decline and the rate of regional atrophy as assessed by MRI scans at baseline and at 24 months across all participants | 24 months
  Clinical decline is assessed by the changes in MMSE (x/30) and CDR (x/3) scores. MRI scans are performed simultaneously during hybrid PET-MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Marie SARAZIN, MD, Prof, Principal Investigator — GHU Sainte-Anne; Guillaume DOROTHEE, PhD, Study Chair — INSERM UMRS 938; Michel BOTTLAENDER, PhD, Study Chair — Service Hospitalier Frédéric Jolit / CEA; Marie Claude POTIER, PhD, Study Chair — Institut du Cerveau et de la Moelle épinière, Hôpital Pitié-Salpêtrière
Locations (3):
- France (3):
  - CHU de Lille, Lille
  - GHU Saint Anne Psychiatrie & Neurosciences, Paris
  - CHU de Rouen, Rouen